CLINICAL TRIAL: NCT02470767
Title: An Observational Cross-sectional Study Evaluating the Sociodemographic and Clinical Characteristics of Patients Diagnosed With NVAF With a Risk of Stroke or Systemic Embolism, Who Are on Treatment to Adequately Control Their Coagulation and Treated in Primary Care Centres
Acronym: SILVER-AP
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17964
Record Dates: First submitted 2015-05-19; First posted 2015-06-12 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Stroke; Prevention and Control; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DOAC treated patients: Patients diagnosed with Non-Valvular Atrial Fribilation at risk of stroke or systemic embolism treated in primary care centres with DOAC.
  Interventions: Drug: Direct Oral Anticoagulant (DOAC)

INTERVENTIONS:
Drug: Direct Oral Anticoagulant (DOAC) — Treatment pattern following the summary of product characteristics

SUMMARY:
describe the sociodemographic and clinical characteristics of patients diagnosed with non-valvular atrial fibrillation (NVAF) at risk of stroke or systemic embolism on anticoagulant therapy who have changed their therapeutic regimen, due to any clinical situation, based on the doctor's routine clinical practice and are currently on treatment with a direct oral anticoagulant (DOAC)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age diagnosed with NVAF with a risk of stroke or systemic embolism treated in primary care centres.
* Patients on regular treatment with anticoagulants who have changed their ther-apeutic regimen due to any clinical situation and have been on treatment with a DOAC for at least three months before being recruited (date of signing the in-formed consent).
* Patients whose DOAC has been indicated by the primary care physician.
* Patients who have given their informed consent in writing.

Exclusion Criteria:

* Patients who changed their anticoagulant therapy within a period of less than three months before signing the informed consent.
* Patients with cognitive impairment preventing them from understanding what is written in the patient information sheet or the informed consent, or from per-forming the self-administered questionnaires.
* Patients who started anticoagulant therapy for NVAF with a DOAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk of stroke or systemic embolism on anticoagulant therapy, who have changed their therapeutic regimen according to their doctor's decision, due to any clinical situation and based on routine clinical practice, and who at the time of enrolment in the study have been receiving treatment with a DOAC for at least three months
Sampling Method: Non-Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Composite of demographic characteristics: age, gender and race | At baseline visit
  sociodemographic data
Composite of relevant cardiovascular events: stroke, TIA, systemic embolism, bleeding | At baseline visit
  clinical characteristics
Composite of comorbidities: hypertension, heart failure, diabetes mellitus, kidney failure, dyslipidemia, | At baseline visit
  clinical characteristics
Data on the Non-Valvular Atrial Fibrillation treatment: relevant active substances | At baseline visit
  clinical characteristics
Concomitant treatments: relevant active substances | At baseline visit
  clinical characteristics
Risk of thromboembolic event based on the CHADS2 score | At baseline visit
  clinical characteristics
Risk of thromboembolic event based on the CHA2DS2-VASc score | At baseline visit
  clinical characteristics
Risk of bleeding based on the HAS-BLED score | At baseline visit
  clinical characteristics

SECONDARY OUTCOMES:
Adherence to treatment | At baseline visit
  use of Haynes-Sackett test
Satisfaction of treatment | At baseline visit
  use of ACTS questionnaire
Reason of the change in treatment: according to Spanish guideline for the SPAF management: IPT (Informe de Posicionamiento Terapeutico) | At baseline visit
  use IPT guideline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain